CLINICAL TRIAL: NCT00314314
Title: A Randomized, Double-Blind Controlled Trial Evaluating the Effect of Intranasal Insulin on Neurocognitive Function in Euthymic Patients With Bipolar Disorder
Brief Title: The Effect of Intranasal Insulin on Neurocognitive Function in Euthymic Patients With Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Roger S. McIntyre, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Insulin
Record Dates: First submitted 2006-04-11; First posted 2006-04-13 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2008-05

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder, memory, executive functioning
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Intranasal Insulin
- 2 (Placebo Comparator)
  Interventions: Drug: Diluent

INTERVENTIONS:
Drug: Intranasal Insulin — Intranasal spray; 40 IU qid; 8 weeks
  Arms: 1
Drug: Diluent — Intranasal spray; 8 weeks
  Arms: 2

SUMMARY:
It is hypothesized that the intranasal administration of insulin will enhance hippocampal-dependent neurocognitive performance in euthymic patients with bipolar I or II disorder. This novel initiative represents a proof-of-concept study that insulin is salient to neurocognitive functioning and deficits in bipolar disorder and represents a novel and safe therapeutic avenue. The available literature suggests that the acute administration of intranasal insulin enhances cognition in memory impaired older adults with either Alzheimer's disease or minimal cognitive impairment. Prior research demonstrates a cognitive enhancing effect of insulin within one hour of the first intranasal insulin dose. Other studies suggest that the long-term administration of intranasal insulin (i.e. over eight weeks) in enhances memory performance in human volunteers. We aim to evaluate the acute and long-term effects of intranasal insulin administration in persons with bipolar disorder. As such we will be conducting the neuropsychological testing at three time points, the week before receiving insulin, within one hour of the first dose and after 8 weeks of insulin administration.

DETAILED DESCRIPTION:
Sixty verified euthymic individuals (age 18-60) with DSM-IV-TR defined Bipolar Disorder (diagnosis will be confirmed by the Mini International Neuropsychiatric Interview for the DSM-IV) will be enrolled. Individuals below the age of 18 and over 60 are excluded as they are not seen at the recruiting center. Enrollment into the study is voluntary. Eligible subjects will provide written informed consent. Subjects will be enrolled from the outpatient Mood Disorders Psychopharmacology Unit (MDPU), University health Network, University of Toronto. Study information and consent procedures will be provided by personnel other than the primary treatment provider.

Euthymia (the absence of clinically meaningful symptoms) will be prospectively defined as a score of 3 or less with the Hamilton Rating Scale for Depression 7 item (HAMD-7) and a score of 7 or less on the Young Mania Rating Scale (YMRS) at initial assessment and at 1 month (baseline). The HAMD-7 and YMRS will be repeated at every follow-up visit.

Conventional pharmacological treatments for bipolar disorder will be permitted (e.g. Lithium, anticonvulsant mood stabilizers, antipsychotics, antidepressants, anxiolytics/hypnotics, etc.). Medication regimens will remain stable throughout the duration of the study. Enrollment into the study is voluntary. Eligible subjects will provide written informed consent. Study information and consent procedures will be provided by personnel other than the primary treatment provider. Subjects will be enrolled from the outpatient Mood Disorders Psychopharmacology Unit, University Health Network, University of Toronto. Illness characteristics will be obtained from the patient interview and hospital medical records.

Subjects will be compensated for sundry expenses (i.e. parking, public transport). Subjects will not receive financial compensation for being a participant in the study. The ongoing provision of care is not contingent on enrollment and/or completion of the study protocol.

Subjects will be excluded if they are receiving corticosteroids or antihypertensive medications; another current Axis I psychiatric disorder; a neurological or medically unstable condition; substance or alcohol misuse in the past 3 months; or electroconvulsive therapy in the last year. Other exclusion criteria include the presence of diabetes mellitus or hyperglycemia, BMI equal or greater than 40 kg/m^2 or inability to provide written informed consent. Patients who are actively suicidal or evaluated as being a suicide risk will be excluded. Other reasons for discontinuation are voluntary discontinuation, failure to complete 1 month of euthymia, impaired fasting glucose (i.e. 6.1-6.9 mmol/L), non-compliance (i.e. failure to administer > 80% of the assigned treatment in any week). Insulin will be measured quantitatively on a weekly basis; subjects will also complete a diary of when they took intranasal insulin and their prescribed medication.

The ongoing provision of care is not contingent on enrollment and/or completion of the study protocol. Furthermore, there will be ongoing communication with the subject's primary care provider in regards to their participation in this study.

This is a randomized double-blind, placebo-controlled, parallel-group study.

The initial visit entails the provision of detailed study information to a subject and obtainment of written informed consent from the subject. The subject will then meet a research team member at a later date for a screening visit. This study requires a total of 12 visits.

Neuropsychological testing will be conducted at 3 time points:

1. Baseline (Visit 3)
2. Within 60 minutes of the first administration of randomized treatment (Visit 4)
3. Endpoint (Visit 12)

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I Disorder - Euthymic
* Bipolar II Disorder - Euthymic

Exclusion Criteria:

* Unstable Medical Conditions
* Currently Manic, Depressed or Mixed

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Cognitive Tests: CVLT, Process Dissociation Tasks | 8 weeks

SECONDARY OUTCOMES:
Cognitive Tests: Trails A | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roger McIntyre, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada